CLINICAL TRIAL: NCT00700557
Title: Lactobacillus Casei e Bifidobacterium Breve as Probiotics at the Treatment of Antibiotic Associated Diarrhea: a Randomized Double Blind Study
Brief Title: Probiotics at the Treatment of Antibiotic Associated Diarrhea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Faculdade de Medicina (FAMED), Agnaldo Coelho da Silva
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: changeme-12332111
Record Dates: First submitted 2008-05-15; First posted 2008-06-18 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Antibiotic-Associated Diarrhea
Keywords: Antibiotic Associated Diarrhea; probiotics; treatment
MeSH Terms: interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotics - Lactobacillus casei and Bifidobacterium breve (Active Comparator): Yakult LB®
  1 sachet (1g) of Lactobacillus casei and Bifidobacterium breve - 6 x 108 UFC/g on a juice three times a day
  Interventions: Dietary Supplement: Probiotics - Lactobacillus casei and Bifidobacterium breve
- maize starch (Placebo Comparator): 725mg on juice three times a day
  Interventions: Dietary Supplement: Maize starch

INTERVENTIONS:
Dietary Supplement: Probiotics - Lactobacillus casei and Bifidobacterium breve — Experimental group:This group received enteral tube feeding or oral diet plus a juice containing 1 sachet (1g) of probiotics (Lactobacillus casei and Bifidobacterium breve - 6x 108 UFC/g) three times a day.
  Arms: Probiotics - Lactobacillus casei and Bifidobacterium breve
Dietary Supplement: Maize starch — Placebo group: This groups received enteral tube feeding or oral diet plus a juice containing,approximately, 725mg of placebo three times a day.
  Arms: maize starch

SUMMARY:
The purpose of this study is to know the efficacy of the treatment with probiotics, Lactobacillus casei and Bifidobacterium breve, on clinical evidences and occurence of relapses on antibiotic-associated diarrhea.

DETAILED DESCRIPTION:
The Antibiotic-Associated Diarrhea (AAD)is defined as that developed after the started antibiotic therapy ou until six to eight weeks after the end of the treatment. The occurence of AAD is about 5% to 25% of the patients using antibiotics and cause watery diarrhea, fever and vomit, mainly on pseudomembranous colitis. Several studies had demonstrated the use of probiotics as therapeutic or preventive form of AAD with or without the presence of C. difficile. About the tolerance of the probiotics,there weren´t observed deleterious effects on health with the consumption of 106 - 107 UFC of Lactobacillus spp and Bifidobacterium spp during a period of one year. The realization of this study can demonstrate the efficacy of Lactobacillus casei e Bifidobacterium breve at the treatment of AAD.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with diarrhea using antibiotic during, at least, 24 hours or had used antibiotic 07 days prior to study entry.

Exclusion Criteria:

* Patients with chronic diarrhea, viral diarrhea, critical patients, during or after radio or chemiotherapy treatment,
* HIV infections,
* Ulcerative colitis,
* Crohn´s disease,
* Hydroelectrolytic disturbance,
* Small intestine syndrome,
* Colostomized, jejunostomized
* Lactose intolerance,
* Rapid enteral diet infusion (>120mh/h),
* Hyperosmolar enteral diet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Reduction of discharge numbers, change the consistency of the feces and occurence of relapses. | After 24 hours of the intervention started

CONTACTS AND LOCATIONS:
Overall Officials: Miguel T Jorge, Medicine, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Federal University of Uberlândia, Uberlândia, Minas Gerais, Brazil